CLINICAL TRIAL: NCT04257799
Title: Lumpectomy Specimen Margin Evaluation With Tomography and Structured Light Imaging
Status: Completed | Type: Observational
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: Trustees of Dartmouth College (Other)
Responsible Party: Principal Investigator, Richard J. Barth,Jr., Chief, Section of General Surgery, Dartmouth-Hitchcock Medical Center
Other Study IDs: D19160
Record Dates: First submitted 2020-02-04; First posted 2020-02-06 (Actual); Last update posted 2022-06-22 (Actual); Status verified 2022-06

CONDITIONS: Breast Cancer Female
MeSH Terms: interventions — Drug Delivery Systems

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Women with breast cancer diagnosis: Women with diagnosis of invasive breast cancer based on pre-surgical biopsy, and scheduled for breast-conserving surgery in the Dartmouth-Hitchcock (DH) Outpatient Surgical Center.
  Interventions: Other: Structured Light Imaging (SLI) System

INTERVENTIONS:
Other: Structured Light Imaging (SLI) System — Investigation of SLI and Tomographic Imaging to see if they will identify cancer cells at the edge of tissue specimens removed during the operation.

SUMMARY:
The purpose of this study is to test a new surgical imaging system called "Structured Light Imaging (SLI)." This system is designed to examine tissue removed during breast cancer surgery to see whether the tissue's edges contain cancer. The current standard of practice is to remove the breast tumor tissue and send the tissue to the lab for analysis following surgery. One in five women (in the US) must later return for a second surgery to remove cancer cells that the lab found remaining in the tissue.

In this study, researchers hope that the new SLI system may detect the cancer cells in the tissue's edges by imaging at the time of surgery. If successful, in the future we may use this system to improve entire cancer removal at the time of surgery, and reduce the need to perform a second surgery to remove additional breast tissue.

DETAILED DESCRIPTION:
On the day of surgery, the surgeon will remove the patient's cancerous tissue, and then in a separate room near the operating room, imaging staff will test it with the Structured Light Imaging system. The testing may take several extra minutes to capture the images. After this imaging, the surgeon will complete the surgery. Following surgery, and per routine medical care, the patient's breast tumor tissue sample will be sent to DHMC's lab for testing. The patient will see her primary doctor for standard surgery follow-up.

No additional imaging or testing will be required for this research study following the usual surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Females 18 years of age or older.
2. Histologic diagnosis of invasive breast cancer based on pre-surgical core biopsy.
3. Scheduled for breast conserving surgery in the Dartmouth-Hitchcock (DH) Outpatient Surgical Center
4. Ability to give an informed consent.

Exclusion Criteria:

1. Patients who will have an expected specimen size greater than the specimen holder (i.e. > 10 X 10 X 5 cm).
2. Prisoners and cognitively impaired adults.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Study Population: The investigators estimate that 100 women will be required. Based on the studies presented in the Introduction, the investigators expect 20% of breast cancer patients to have a positive margin.
  Based on historical operative volumes, the investigators anticipate recruiting 2 breast cancer patients per week. Thus it will take one year to accrue 100 patients to the study.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2020-02-06 (Actual); Primary Completion 2022-03-16 (Actual); Study Completion 2022-03-16 (Actual)

PRIMARY OUTCOMES:
Sensitivity and Specificity of 3D tomography-SLI as measured by concurrence with standard of care 2-D mammography | Day of surgery
  Two surfaces (anterior and posterior) will be evaluated by SLI and 6 surfaces (anterior, posterior, medial, lateral, cranial, and caudal) will be evaluated by 3D tomography. Four surfaces are evaluated by standard-of-care 2-dimensional specimen mammography: medial, lateral, cranial and caudal to evaluate for the presence of cancer at the margin. Since anterior and posterior surfaces will be evaluated by both 3D tomography and SLI, an anterior or posterior margin will be considered positive only if it is positive by both 3D tomography and SLI. Otherwise the margin will be considered negative.
  Sensitivity will be computed as True Positive (TP)/TP + False Negative (FN) results, compared to pathology. Specificity will be computed as True Negative (TN)/TN + False Positive (FP) results, compared to pathology.

SECONDARY OUTCOMES:
Sensitivity and Specificity of 3D tomography alone in identifying true positive margins and true negative margins | Day of Surgery
  Sensitivity will be computed as True Positive (TP)/TP + False Negative (FN) results compared to pathology. Specificity will be computed as True Negative (TN)/TN + False Positive (FP) results compared to pathology.
Sensitivity and Specificity of SLI alone in identifying true positive margins and true negative margins | Day of Surgery
  Sensitivity will be computed as True Positive (TP)/TP + False Negative (FN) results compared to pathology. Specificity will be computed as True Negative (TN)/TN + False Positive (FP) results compared to pathology.
Sensitivity and Specificity of standard-of-care 2D specimen mammography | Day of Surgery
  The investigators will calculate the sensitivity and specificity of standard-of-care 2D specimen mammography and compare that to the combination of 3D tomography and SLI. Sensitivity will be computed as TP/TP + FN results compared to pathology. Specificity will be computed as TN/TN + FP results compared to pathology.
Determine the logistics of use of the imaging system, software interface and specimen holder. | Day of Surgery
  The investigators will determine the logistics of use of the imaging system, software interface and specimen holder for possible future refinement.

CONTACTS AND LOCATIONS:
Overall Officials: Richard J Barth Jr., MD, Principal Investigator — DHMC
Locations (1):
- Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No